CLINICAL TRIAL: NCT01140984
Title: An Investigator Initiated Open Study to Evaluate the Efficacy and Safety of Intra Arterial Infusion for Treatment of Steroid Resistant Acute Hepatic Graft Versus Host Disease (AGVHD)
Brief Title: Intra Arterial (IA) Steroids Infusion for Hepatic Acute Hepatic Graft Versus Host Disease (aGVHD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: technical issues
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYS-08-HMO-CTIL
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2011-02

CONDITIONS: Acute Graft Versus Host Disease
Keywords: acute graft versus host disease; intra arterial steroid infusion; steroid resistant acute hepatic graft versus host disease
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: Methylprednisolone (Intra-arterial continuous infusion of corticosteroids)

INTERVENTIONS:
Drug: Methylprednisolone (Intra-arterial continuous infusion of corticosteroids) — Sedation/anesthesia of patient followed by placement of a 4F vascular sheath and a diagnostic and hepatic angiogram. Angiographic catheter tip to be placed in the proximal proper hepatic artery, secured in place externally and connected to an arterial line pressurized system which allows continuous drip infusion of methylprednisolone diluted in normal saline (600mg/m2 with maximal total dose of 100mg diluted in 480cc in normal saline administered at 20cc/hr for 24 hours).

SUMMARY:
Post allogeneic hematopoietic stem cell transplantation (HSCT) patients with steroid resistant acute GVHD localised to the liver will receive 24 hours continuous intra-arterial infusion of methylprednisolone.

DETAILED DESCRIPTION:
The study population will include 30 patients with SR AGVHD having an index of B, C, or D on the IBMTR severity index localized to the liver.

Standard treatment for SR AGVHD includes: IV cyclosporine or tacrolimus with adjusted doses depending on serum levels and methylprednisolone or prednisone 2 mg/kg/d. This treatment may be continued during the study period although steroid taper down should be attempted if clinically possible.

GVHD diagnosis will be based upon clinical criteria and biopsy (if needed) from an involved organ. GVHD will be graded according to the International Bone Marrow Transplantation Registry (IBMTR) severity index.

Intra-arterial treatment should be given in less than 72h from completion of inclusion criteria.

Partially responding or non-responding patients may receive a second treatment within 14 days of the initial intra-arterial treatment, at the discretion of the treating physician.

Definitions

Hepatic response:

* Initial response - the day in which bilirubin level began to decrease.
* Partial response 75 - the day in which bilirubin level decreased below 75% of basal level.
* Partial response 50 - the day in which bilirubin level decreased below 50% of basal level.
* Partial response 25 - the day in which bilirubin level decreased below 25% of basal level.
* Complete response - the day in which bilirubin level decreased to normal level.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of allogeneic stem cell transplantation.
* Age>18 years.
* Post stem cells transplant <100 days.
* AGVHD of liver, IBMTR index B, C, D.
* Resistant AGVHD - Patients will be eligible for inclusion if they developed grade B-D AGVHD with progression after 3 days standard treatment OR unresponsive to at least 7 days standard treatment OR incomplete response to standard treatment after 14 days.
* Has received no 1st line treatment for steroid refractory AGVHD.
* Signed a written informed consent

Exclusion Criteria:

* Not fulfilling any of the inclusion criteria.
* Active life-threatening infection.
* Inability to comply with study requirements.
* Inability to give informed consent.
* Contraindication to arterial catheterization (uncorrectable coagulopathy, severe allergic reaction to contrast material or others).
* Inability to give the first Intra-arterial treatment in less than 72h from completion of inclusion criteria
* An IBMTR index ≤ A.
* Refractory skin AGVHD or severe diarrhea..
* Pregnant or breast-feeding female or childbearing potential.
* Known to be HIV positive.
* Has been diagnosed with veno-occlusive disease.
* Has been diagnosed with multi organ failure.
* Known renal failure eGFR <30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Hepatic response | 180 days
  The degree to which serum bilirubin levels do or do not decrease

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organisation, Jerusalem, Israel

REFERENCES:
- [Background] Billaud EM. Clinical pharmacology of immunosuppressive drugs: year 2000--time for alternatives. Therapie. 2000 Jan-Feb;55(1):177-83. PMID 10860022
- [Background] Tanner JE, Alfieri C. Interactions involving cyclosporine A, interleukin-6, and Epstein-Barr virus lead to the promotion of B-cell lymphoproliferative disease. Leuk Lymphoma. 1996 May;21(5-6):379-90. doi: 10.3109/10428199609093435. PMID 9172802
- [Background] Brandenburg U, Gottlieb D, Bradstock K. Antileukemic effects of rapid cyclosporin withdrawal in patients with relapsed chronic myeloid leukemia after allogeneic bone marrow transplantation. Leuk Lymphoma. 1998 Nov;31(5-6):545-50. doi: 10.3109/10428199809057613. PMID 9922044
- [Background] Graziani F, Van Lint MT, Dominietto A, Raiola AM, Di Grazia C, Lamparelli T, Gualandi F, Bregante S, Fiorone M, Bruno B, Bacigalupo A. Treatment of acute graft versus host disease with low dose-alternate day anti-thymocyte globulin. Haematologica. 2002 Sep;87(9):973-8. PMID 12217810
- [Background] MacMillan ML, Weisdorf DJ, Davies SM, DeFor TE, Burns LJ, Ramsay NK, Wagner JE, Blazar BR. Early antithymocyte globulin therapy improves survival in patients with steroid-resistant acute graft-versus-host disease. Biol Blood Marrow Transplant. 2002;8(1):40-6. doi: 10.1053/bbmt.2002.v8.pm11858189.
- [Background] Tagliabue A, Corti P, Vigano E, Bonanomi S, Uderzo C. Favourable response to antithymocyte globulin therapy in resistant acute graft-versus-host disease. Bone Marrow Transplant. 2005 Sep;36(5):459. doi: 10.1038/sj.bmt.1705065. No abstract available. PMID 15980883
- [Background] Arai S, Margolis J, Zahurak M, Anders V, Vogelsang GB. Poor outcome in steroid-refractory graft-versus-host disease with antithymocyte globulin treatment. Biol Blood Marrow Transplant. 2002;8(3):155-60. doi: 10.1053/bbmt.2002.v8.pm11939605.
- [Background] Khoury H, Kashyap A, Adkins DR, Brown RA, Miller G, Vij R, Westervelt P, Trinkaus K, Goodnough LT, Hayashi RJ, Parker P, Forman SJ, DiPersio JF. Treatment of steroid-resistant acute graft-versus-host disease with anti-thymocyte globulin. Bone Marrow Transplant. 2001 May;27(10):1059-64. doi: 10.1038/sj.bmt.1703032. PMID 11438821
- [Background] Roy J, McGlave PB, Filipovich AH, Miller WJ, Blazar BR, Ramsay NK, Kersey JH, Weisdorf DJ. Acute graft-versus-host disease following unrelated donor marrow transplantation: failure of conventional therapy. Bone Marrow Transplant. 1992 Jul;10(1):77-82. PMID 1515883
- [Background] Weisdorf D, Haake R, Blazar B, Miller W, McGlave P, Ramsay N, Kersey J, Filipovich A. Treatment of moderate/severe acute graft-versus-host disease after allogeneic bone marrow transplantation: an analysis of clinical risk features and outcome. Blood. 1990 Feb 15;75(4):1024-30. PMID 2302454
- [Background] Martin PJ, Schoch G, Fisher L, Byers V, Appelbaum FR, McDonald GB, Storb R, Hansen JA. A retrospective analysis of therapy for acute graft-versus-host disease: secondary treatment. Blood. 1991 Apr 15;77(8):1821-8. PMID 2015405
- [Background] Bloom AI, Shapira MY, Or R, Sasson T, Resnick IB, Zilberman I, Verstandig A, Aker M, Slavin S, Muszkat M. Intrahepatic arterial administration of low-dose methotrexate in patients with severe hepatic graft-versus-host disease: an open-label, uncontrolled trial. Clin Ther. 2004 Mar;26(3):407-14. doi: 10.1016/s0149-2918(04)90036-7. PMID 15110133
- [Background] Sato T, Sakamaki S, Nagaoka Y, Kuribayashi K, Nagamachi Y, Morii K, Honma H, Kogawa K, Kato J, Niitsu Y. Intra-mesenteric artery steroid administration relieved severe refractory gastro-intestinal graft-vs.-host disease in an allogeneic bone marrow transplantation patient. Am J Hematol. 1997 Dec;56(4):277-80. doi: 10.1002/(sici)1096-8652(199712)56:43.0.co;2-6. PMID 9395192
- [Background] Nakai K, Tajima K, Tanigawa N, Matsumoto N, Zen K, Nomura S, Fujimoto M, Kishimoto Y, Amakawa R, Sawada S, Fukuhara S. Intra-arterial steroid-injection therapy for steroid-refractory acute graft-versus-host disease with the evaluation of angiography. Bone Marrow Transplant. 2004 Jun;33(12):1231-3. doi: 10.1038/sj.bmt.1704523. PMID 15094752